CLINICAL TRIAL: NCT05859282
Title: Development and Validation of a Short Tool to Assess the Awareness of Pregnancy-induced Hypertension: A Cross-sectional Study Among Pregnant Women in Lebanon
Brief Title: Development and Validation of a Short Tool to Assess the Awareness of Pregnancy-induced Hypertension
Status: Completed | Type: Observational
Sponsor: Georges Hatem (Other)
Responsible Party: Sponsor-Investigator, Georges Hatem, Sponsor-Principal investigator, Lebanese University
Organization: Lebanese University (Other)
Other Study IDs: 2D/21/10
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy Related; Hypertension in Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Survey — A short 25-item tool was developed and can be applied in clinics to assess the awareness of pregnancy hypertension.

SUMMARY:
Background: Pregnancy-induced hypertension (PIH) is responsible for most perinatal and fetal mortality. Few programs are patient-centered during pregnancy, increasing the risks of misinformation and misconceptions among pregnant women and, as a result, malpractices. Objective: This study aims to develop and validate a form to assess the knowledge and attitudes of pregnant women about PIH.

DETAILED DESCRIPTION:
Many observational studies explored the awareness of pregnant women of PIH, but no structured tool is available to assess such awareness. During the past two years, education campaigns were postponed and primary care was prioritized. To allow better-informed decisions and targeted actions, this pilot study aims to develop and validate a short form to assess the knowledge and attitudes of pregnant women about pregnancy-induced hypertension. The long-term objective of this study is to provide a practical tool for pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Participants were asked to participate in the study with no criteria based on race, ethnicity, or gestational age.

Exclusion Criteria:

* Those with a history of hypertension or pre-eclampsia were excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women were targeted from five obstetrics and gynecology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-11-07 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Awareness of hypertensive disorders of pregnancy by developing a 25-item questionnaire | 6 months
  Thirty-six statements were initially provided to which women had to answer either ''yes'', ''No'' or ''I don't Know''. Out of these statements, 25 were retained due to positive inter-item correlation (15 knowledge statements and 10 behavior statements), and the other statements were eliminated one by one after testing for reliability and computing the effect of each statement on the internal consistency.

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese University Faculty of pharmacy, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided